CLINICAL TRIAL: NCT03209375
Title: Identification of the Sick Patient in the ED
Status: Completed | Type: Observational
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 217746
Record Dates: First submitted 2017-06-28; First posted 2017-07-06 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Emergencies
Keywords: triage; early warning system
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional study will test scoring systems used to identify high risk patients when they are triaged upon presentation in the Emergency Department (ED) in a single hospital in the Northwest of England between May and July 2017.E The study will involve collecting data only from a cohort of 500 consecutive patients who arrive at the ED. Patients who have a traumatic, purely obstetric or purely psychiatric condition will be excluded.

Patients will be triaged as is routine by nursing and medical staff using various scoring methods determine whether they are high risk and need urgent, life-saving treatment. In addition the impression (yes/no) of the triaging nurse and the treating clinician as to whether the patient will need a life-saving intervention will be collected. Patients will be followed up for 48 hours to see whether they needed any life-saving treatment, such as admission to ICU, life-saving surgery, cardiopulmonary resuscitation (CPR), or death.

Each patient's Manchester Triage category, NEWS at presentation, nurse and treating clinician impressions and a novel score calculated from NEWS data will be collected together with the outcome data in order to compare the predictive power of the five scoring systems. In this way the study will test which is the best scoring system for identifying high risk patients in a timely manner. This is important as it can allow life saving treatment to be delivered quickly to those patients who need it most and can prevent inappropriate interventions on patients who do not immediately need them. The study will collect minimal patient information and will not interfere with or alter their treatment in any way. Only patient data recorded as part of routine practice is required, which will be collected by members of the direct care team and will be anonymised prior to analysis.

DETAILED DESCRIPTION:
This is a single-centre, non-interventional, prospective observational cohort study collecting data from patients presenting to the ED of a large teaching hospital in the Northwest of England. The study is designed to gather information about the number of patients receiving life-saving intervention within 48 hours of presentation and the best of five proposed ways of identifying these patients when they present to the ED. This study is non-interventional and there will be no interference with treatment decisions or alteration in clinical practice.

A prospective observational approach is chosen as it will allow direct access to information and better capture of the systems being assessed in the ED. Information about each patient's perceived risk at presentation (in terms of the five proposed systems) will be collected at the time of presentation. Information will include rating on the five proposed systems and a number of outcome variables, all of which are recorded as part of routine clinical practice. All information will be captured directly into a specially designed database including a study number to preclude the need to record any personal identifiable information for the study.

Data will be collected for each patient on an anonymised database. Demographic details (age, gender, presenting condition) will be collected to identify if the sample is representative of a general ED population. Each patient's Manchester Triage category, NEWS at presentation and the novel score calculated from NEWS data will be included, as will the impression (yes/no) of the triaging nurse and the treating clinician as to whether the patient will need a lifesaving intervention. A number of outcome measures (death, admission to high dependency or intensive care, admission directly to the cardiac catheter laboratory or coronary care, emergency endoscopy, thrombolysis, life-saving surgery, intubation, emergency intravenous medication, CPR, DC cardioversion/external or internal cardiac pacing, massive transfusion for ongoing haemorrhage and non-invasive ventilatory support) will be extracted, having been defined a priori as being potentially life-saving. The demographic details and variables chosen are all recorded or calculated for each patient as part of routine practice on critical care. No additional tests or measurements will be required for this study.

Data will be anonymised by allocation of a study number and this figure will be cross-referenced to an electronic masterlist which will contain the patient name and hospital number. In this way the database can be linked back to the patient to continue data collection and entry. The masterlist will be an electronic spreadsheet which will be stored on a secure server at the hospital and accessed via password protected computers within the ED. The masterlist will be destroyed on completion of the study.

Patient information will be collected in a spreadsheet designed to collate the information and allow statistical analysis. No identifiable patient information will be inputted onto the spreadsheet

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Royal Preston Hospital Emergency Department

Exclusion Criteria:

* Trauma, purely psychiatric or obstetric presentation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As above.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Life-saving intervention | 48 hours
  Composite outcome measure

SECONDARY OUTCOMES:
Death | 48 hours
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Challen, PhD, Principal Investigator — Lancashire Teaching Hospital NHS Trust
Locations (1):
- Royal Preston Hospital, Preston, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided